CLINICAL TRIAL: NCT03615846
Title: Comparison of the VerifyNow® Aspirin Test and PRUTest® Platelet Reactivity Tests With Investigational Reagent to Reagents Registered in Japan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Accriva Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: VFN-CSS-19-0008
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Platelet Aggregation; Coronary Artery Disease
Keywords: Platelet Aggregation; P2Y12 Inhibitor
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dual Anti-Platelet Therapy (DAPT): Whole blood from patients who are currently receiving Dual Anti-Platelet Therapy (DAPT) Clopidogrel and aspirin (ASA) for a minimum of 4 weeks (on-drug) will be used to conduct antiplatelet reactivity tests using VerifyNow assay and LTA with AggRAM Aggregometer with and without PGE1.
  There is no drug administration or therapeutic intervention in this study. The results of platelet activation testing using VerifyNow performed in this study are not used to influence patient care.
- One Anti Platelet Medication Only: Whole blood from patients who are currently receiving either ASA or Clopidogrel alone for a minimum of 4 weeks (on-drug) will be used to conduct antiplatelet reactivity tests using VerifyNow assay and LTA with AggRAM Aggregometer with and without PGE1.
  There is no drug administration or therapeutic intervention in this study. The results of platelet activation testing using VerifyNow performed in this study are not used to influence patient care.
- naive: No medication with anti-platelet effects There is no drug administration or therapeutic intervention in this study. The results of platelet activation testing using VerifyNow performed in this study are not used to influence patient care.

SUMMARY:
This is a multi-center convenience sample prospective study comparing the results of the Verify Now® Aspirin Test and PRUTest® Platelet Reactivity Tests with the Japan investigational reagents to reagents registered in Japan in the expected population receiving aspirin (ASA) and the P2Y12 inhibitor clopidogrel.

DETAILED DESCRIPTION:
* The Primary Objectives of this study are to compare the results of:
* The VerifyNow Aspirin Test with AA, an investigational reagent as defined in Japan, against LTA with AA investigational reagent as defined in Japan (study reference reagent), in subjects receiving DAPT (ASA and clopidogrel or subjects taking no platelet inhibitors including ASA;
* The VerifyNow Aspirin Test with AA, an investigational reagent as defined in Japan, against LTA with collagen (study reference reagent),

  o In subjects receiving DAPT (ASA and clopidogrel) or in subjects taking no platelet inhibitors including ASA
* The VerifyNow PRUTest with ADP, an investigational reagent as defined in Japan, and PGE1, against LTA with ADP, an approved reagent in Japan (study reference reagent) and PGE1, and
* The VerifyNow PRUTest with ADP (an investigational reagent as defined in Japan) and PGE1 against LTA with ADP reagent approved in Japan (study reference reagent) with no PGE1, o in up to 75 subjects receiving DAPT (ASA and clopidogrel) and in up to 55 subjects taking no platelet inhibitors (total up to 130 subjects).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age or older.
* Subjects regularly taking ASA and clopidogrel, for a minimum of 4 days prior to enrollment, or subjects taking no platelet inhibitors including ASA.
* Willing to participate and able to understand the study, including their rights and any risks associated with their participation, and sign an informed consent.
* Able and willing to donate a blood sample of 15mL.

  • Exclusion Criteria
* Enrolled in any other study that involves an investigational drug and/or device.
* Smoked within one hour before blood draw.
* Had caffeine within 2 hours before blood draw.
* Had meals with high fat content within 8 hours before blood draw.
* A platelet count below 92,000/µL, or above 502,000/µL for VerifyNow Aspirin Test.*
* A platelet count below 119,000/µL, or above 502,00/µL for VerifyNow PRUTest.*
* A hematocrit level below 29%, or above 56% for VerifyNow Aspirin Test.*
* A hematocrit level below 33%, or above 52% for VerifyNow PRUTest.*
* Within the past 48 hours, exposure to any of the following drugs:

  * Antiplatelet/glycoprotein inhibitors [eptifibatide, tirofiban]
  * Any antiplatelet drug except clopidogrel and ASA [e.g. ticagrelor, prasugrel]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population to be studied consists of subjects who are currently receiving Dual Anti-Platelet Therapy (DAPT) Clopidogrel and aspirin (ASA) or receiving either ASA or Clopidogrel alone for a minimum of 4 weeks, or subjects receiving no drugs with anti-platelet effect.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
VerifyNow® PRUTest | 1 day
  Correlation of AggRAM Light Transmittance Aggregometry (LTA) compared to VerifyNow PRUTest
VerifyNow® Aspirin Test | 1 day
  Correlation of AggRAM Light Transmittance Aggregometry (LTA) compared to VerifyNow Aspirin Test
Naive | 1 day
  Correlation of AggRAM Light Transmittance Aggregometry (LTA) compared to VerifyNow Aspirin Test and VerifyNow PRUTest

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rubinstein, MD, Study Chair — Instrumentation Laboratory; Michael Martin, Study Director — Accrira Diagnostics / Instrumentation Laboratory
Locations (2):
- United States (2):
  - Accriva Study Site, Jacksonville, Florida
  - Accriva Study Site, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No